CLINICAL TRIAL: NCT01067131
Title: A Phase I Randomized Placebo Controlled Study of a Virosome Formulated Anti-Candida Vaccine (PEV7) Administered by the Vaginal (PEV7C) or Intramuscular (PEV7B) Route to Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity Study of a Virosomal Vaccine Against Recurrent Vulvovaginal Candida Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pevion Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PCAN001
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Vulvovaginal Candidiasis
Keywords: Candida albicans; Fungal vaginal infection; Vulvovaginal candidiasis; Candidose; Vaccine; Virosome
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PEV7C1, intravaginal (Experimental): Vaccine containing virosomes intravaginally applied
  Interventions: Biological: PEV7C1
- PEV7C9, placebo, intravaginal (Placebo Comparator): Placebo vaccine (excipient only) intravaginally applied
  Interventions: Biological: PEV7C9
- PEV7B2, intramuscular low dose (Experimental): Intramuscular vaccine low dose of antigen
  Interventions: Biological: PEV7B2
- PEV7B1, intramuscular high dose (Experimental): Intramuscular vaccine, high dose of antigen
  Interventions: Biological: PEV7B1

INTERVENTIONS:
Biological: PEV7C1 — capsule intravaginal application contains antigen coupled to virosomes
  Arms: PEV7C1, intravaginal
Biological: PEV7C9 — capsule intravaginal application contains excipient only
  Arms: PEV7C9, placebo, intravaginal
Biological: PEV7B2 — reconstituted lyophilisate intramuscular application contains antigen at low dose coupled to virosomes
  Arms: PEV7B2, intramuscular low dose
Biological: PEV7B1 — reconstituted lyophilisate intramuscular application contains antigen at high dose coupled to virosomes
  Arms: PEV7B1, intramuscular high dose

SUMMARY:
Pevion Biotech develops a state-of-the-art vaccine against recurrent vulvovaginal candidiasis (RVVC) caused by the pathogenic form of Candida albicans especially in pre-menopausal women of childbearing age with a history of recurrent vulvovaginal candidiasis. This study is designed to evaluate the safety and tolerability of the vaccine, administered by two different routes (intramuscular and intravaginal) as primary endpoint. Immunogenicity will be evaluated as secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 45 years.
* Written informed consent obtained from the volunteer.
* Free of obvious health problems as established by medical history and/or clinical examination and/or gynecological examination before entering the study.
* Body Mass Index between 18.0 and 30.0.
* A negative pregnancy test and an adequate contraception until at least 4 weeks after the last vaccination of the primary vaccination course. Adequate contraception means use of a physician-prescribed oral hormonal agent AND use of condoms (without spermicidal agents) at the same time. Progesterone-only contraceptives are not suitable due to the lack of a regular menstrual cycle.
* Availability for the duration of the study and willingness to attend all scheduled visits.
* No vaginal practices other than receptive intercourse with male or use of sanitary tampons during menses.
* Negative culture for any Candida species before visit 2. Subjects with a positive culture will be treated and the Candida culture will be repeated. They will be eligible if a negative culture result is available prior to visit 2 (first vaccination).

Exclusion Criteria:

* Known or suspect history of cervico-vaginal malignancy or abnormality discovered at time of screening. Ovarectomised and hysterectomised women are excluded from the study.
* Presence of Chlamydia trachomatis, Neisseria gonorrhoeae infection as detected by PCR at screening visit.
* Presence of bacterial vaginosis (assessed by the Amsel criteria and bacterial culture) for group 1 and 2 at screening visit; at days 0±2, 28±2 and 56±2, for group 3 and 4 at screening and by Amsel criteria only at days 0±2 and 28±2.
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period and safety follow-up.
* Planned use of any registered vaccine other than study vaccine and planned use of immunoglobulin-based therapy during the immunization phase until 14 days after the last immunization (Day 0 to day 70 for group 1 and 2; Day 0 to Day 56 for group 3 and 4) and for groups 1 and 2 from application of booster vaccine dose until 14 days after administration.
* Receipt of live attenuated vaccine within 30 days prior to the first vaccination until 30 days after the last vaccination of the immunization period. Equally the above applies to the period 30 days prior until 30 days after the booster vaccination.
* Any therapy or medications via vaginal route 7 days prior to first vaccination and in the period from first dose of study vaccine until the last safety visit (Groups 1 and 2: Day 140±2; Groups 3 and 4: Day 70±2). Equally the above applies to the period 7 days prior to booster vaccination until end of study (Groups 1 and 2).
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this will mean prednisone, or equivalent, > 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Samples obtained at screening visit show:

  1. a clinically significant amount of protein and/or haemoglobin in the urine sample
  2. a clinically significant abnormality in the haematological or biochemicals assays
  3. positive antibody assays for Hepatitis B and/or C and/or HIV
* Any chronic drug therapy to be continued during the study period (except oral hormonal contraceptives)
* Any confirmed or suspected acquired immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, or history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine or component used during the manufacturing process of the vaccine like eggs and chick proteins.
* Acute disease at the time of enrollment. {Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., temperature <38°C (<100.4°F)}.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, blood disorder or immune dysfunction as determined by physical examination or laboratory screening tests.
* Acute or chronic diabetes.
* History of chronic alcohol consumption and/or intravenous drug abuse.
* Pregnancy or lactation.
* Subject planning to become pregnant.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Systemic and local AE rates / SAE rates | Immunization period + 3 months

SECONDARY OUTCOMES:
Titers of vaccine antigen specific antibodies | Immunisation phase, last immunisation +2 weeks, +1 month, +3 months, +6 months, +12 months, +14 months (Groups 1&2 only), +15 months (Groups 1&2 only)
Neutralisation capacity of vaccine antigen specific antibodies | Immunisation phase, last immunisation +2 weeks, +1 month, +3 months, +6 months, +12 months, +14 months (Groups 1&2 only), +15 months (Groups 1&2 only)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, Prof, Principal Investigator — Centre hospitalier universitaire vaudois, Vaccine and Immunotherapy Center; Rolf Pokorny, MD, MSc, Principal Investigator — Covance Clinical Research Unit AG
Locations (2):
- Switzerland (2):
  - Covance Clinical Research Unit AG, Allschwil, Basel
  - CHUV, Vaccine and Immunotherapy Center, Lausanne